CLINICAL TRIAL: NCT04465812
Title: The Impact of a Smartphone-based Self-monitoring and Personalized Feedback Multiple Intervention on Cognitive and Cerebrovascular Health in CIRCLE-CHINA
Brief Title: The Impact of a Smartphone-based Personalized Intervention on Cognitive and Cerebrovascular Health in CIRCLE-CHINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing Gaobu Street Community Health Service Center (Unknown); Shaoxing Mashan Street Community Health Service Center (Unknown); Shaoxing Doumen Street Community Health Service Center (Unknown)
Responsible Party: Principal Investigator, Min Lou, Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIRCLE-CHINA II
Record Dates: First submitted 2020-06-28; First posted 2020-07-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Impairment; Stroke; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard health counseling at baseline (No Intervention): Standard health counseling at baseline
- Self-monitoring and personalized feedback on smartphone app (Experimental): 1. Patients will record their blood pressure (once 1-week for patients with hypertension, every 3-month for those without), blood glucose (once 1-month for patients with diabetes), serum lipid metabolism (every 3-month for patients with dyslipidemia) on app, and medical staff will suggest continuing monitoring and recording or recommend outpatient visit;
  2. Patients will complete Pittsburgh sleep quality index test on app every 3-month, and medical staff will contact with patients with index > 15 to assess detail clinical status and recommend outpatient visit if necessary;
  3. Patients will complete Self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS) on app every 3-month, and medical staff will contact with patients with SAS>49 or SDS>52 to assess detail clinical status and recommend outpatient visit if necessary;
  4. Patients will complete cognitive training games every week on app;
  5. Medical staff will send health information on app
  Interventions: Behavioral: Self-monitoring and personalized feedback on smartphone app

INTERVENTIONS:
Behavioral: Self-monitoring and personalized feedback on smartphone app — 1. Patients will record their blood pressure (once 1-week for patients with hypertension, every 3-month for those without), blood glucose (once 1-month for patients with diabetes), serum lipid metabolism (every 3-month for patients with dyslipidemia) on app, and medical staff will suggest continuing monitoring and recording or recommend outpatient visit;
  2. Patients will complete Pittsburgh sleep quality index test on app every 3-month, and medical staff will contact with patients with index > 15 to assess detail clinical status and recommend outpatient visit if necessary;
  3. Patients will complete Self-Rating Anxiety Scale (SAS) and Self-Rating Depression Scale (SDS) on app every 3-month, and medical staff will contact with patients with SAS>49 or SDS>52 to assess detail clinical status and recommend outpatient visit if necessary;
  4. Patients will complete cognitive training games every week on app;
  5. Medical staff will send health information on app
  Arms: Self-monitoring and personalized feedback on smartphone app

SUMMARY:
This smartphone-based personalized multiple intervention study aims to prevent cognitive impairment and reduce dementia and cerebrovascular events in 45-74 year old persons with high risk of stroke in China. The investigators plan to monitor and manage participants' behavioral and health (vascular risk factors control, sleep quality, mental health and cognitive training) based on self-monitoring and personalized feedback via smartphone app. The short-term primary outcome is 1-year change in global cognitive score measured by a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol. The investigators hypothesize that the intervention based on self-monitoring and personalized feedback will prevent cognitive decline by the initial 1-year intervention. The long-term primary outcome is the development of dementia and cerebrovascular events during a total of 5 years' follow-up. The investigators hypothesize that the smartphone-based personalized multiple intervention may reduce the 5-year risk of dementia and cerebrovascular events, mainly through the improvement in vascular risk factors control, sleep quality, mental health and cognitive training activities.

DETAILED DESCRIPTION:
Patients with ≥ 3 stroke risk factors (including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke), or with transient ischemic attack, are regarded as patients with high risk of stroke. Studies have indicated that these stroke risk factors might be associated with an increased risk of cerebral small vessel disease (CSVD) progress, glymphatic dysfunction, cognitive decline, dementia, and cerebrovascular events. However, prevention in these patients is largely unknown and the management of these patients is a very troublesome issue. Previous study has demonstrated that interventions in the feedback and monitoring method could improve exercise adherence in older people compared with other methods including comparison of behavior, social support, natural consequences, identity and goals and planning. Therefore, the investigators plan to monitor and manage vascular risk factors control, sleep quality, mental health and cognitive training based on self-monitoring and personalized feedback on a smartphone app in patients with high risk of stroke. The investigators hypothesize that the intervention based on self-monitoring and personalized feedback will reduce cognitive impairment, glymphatic dysfunction, CSVD progress, depressive symptoms, anxious symptoms, improve sleep quality, and reduce dementia and cerebrovascular events incidence in the study group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* aged 45-74 years
* high risk of stroke (with ≥ 3 of 8 stroke risk factors, including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke, or with transient ischemic attack)

Exclusion Criteria:

* previously diagnosed dementia
* previously diagnosed stroke (both cerebral infarction and hemorrhage)
* suspected dementia after clinical assessment by study physician at screening visit
* disorders affecting safe engagement in the intervention (eg, malignant disease, major depression, symptomatic cardiovascular disease, revascularisation within 1 year previously)
* severe loss of vision, hearing, or communicative ability;
* disorders preventing cooperation as judged by the study physician
* coincident participation in another intervention trial
* any MRI contraindications

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol | 1 year
  Primary Outcome

SECONDARY OUTCOMES:
The change of cognitive score for each domain of NINDS-CSN battery from baseline to 12-month（attention, executive, Language, visuomotor speed, visuospatial function, memory） | 1year
  Short-term Secondary Outcome
Cognitive function change assessed by scores of Mini-Mental State Examination (MMSE) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 1 year
  Short-term Secondary Outcome
Cognitive function change assessed by scores of Montreal Cognitive Assessment (MoCA) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 1 year
  Short-term Secondary Outcome
Dementia and cerebrovascular events incidence | 1 year
  Short-term Secondary Outcome
Changes in glymphatic function assessed by dispersion coefficient of periarterial and perivenous spaces on DTI | 1 year
  Short-term Secondary Outcome
Changes in image markers (WMHs, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 1 year
  Short-term Secondary Outcome
Dementia and cerebrovascular events incidence | 5 years
  Long-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton depression scale (HAMD) (minimum value = 0, maximum value = 77, and higher scores mean a worse outcome) | 1 year
  Short-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton anxiety scale (HAMA) (minimum value = 0, maximum value = 56, and higher scores mean a worse outcome) | 1 year
  Short-term Secondary Outcome
Sleep quality assessed by Pittsburgh sleep quality index (minimum value = 0, maximum value = 21, and higher scores mean a worse outcome) | 1 year
  Short-term Secondary Outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol | 5 years
  Long-term Secondary Outcome
Cognitive function change assessed by scores of Mini-Mental State Examination (MMSE) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  Long-term Secondary Outcome
Cognitive function change assessed by scores of Montreal Cognitive Assessment (MoCA) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  Long-term Secondary Outcome
Changes in image markers (WMHs, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 5 years
  Long-term Secondary Outcome
Changes in glymphatic function assessed by dispersion coefficient of periarterial and perivenous spaces on DTI | 5 years
  Long-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton depression scale (HAMD) (minimum value = 0, maximum value = 77, and higher scores mean a worse outcome) | 5 years
  Long-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton anxiety scale (HAMA) (minimum value = 0, maximum value = 56, and higher scores mean a worse outcome) | 5 years
  Long-term Secondary Outcome
Sleep quality assessed by Pittsburgh sleep quality index (minimum value = 0, maximum value = 21, and higher scores mean a worse outcome) | 5 years
  Long-term Secondary Outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol | 2 years
  Long-term Secondary Outcome
Dementia and cerebrovascular events incidence | 2 years
  Long-term Secondary Outcome
Cognitive function change assessed by scores of Mini-Mental State Examination (MMSE) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  Long-term Secondary Outcome
Cognitive function change assessed by scores of Montreal Cognitive Assessment (MoCA) (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  Long-term Secondary Outcome
Changes in image markers (WMHs, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 2 years
  Long-term Secondary Outcome
Changes in glymphatic function assessed by dispersion coefficient of periarterial and perivenous spaces on DTI | 2 years
  Long-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton depression scale (HAMD) (minimum value = 0, maximum value = 77, and higher scores mean a worse outcome) | 2 years
  Long-term Secondary Outcome
Depressive symptoms assessed by scores of Hamilton anxiety scale (HAMA) (minimum value = 0, maximum value = 56, and higher scores mean a worse outcome) | 2 years
  Long-term Secondary Outcome
Sleep quality assessed by Pittsburgh sleep quality index (minimum value = 0, maximum value = 21, and higher scores mean a worse outcome) | 2 years
  Long-term Secondary Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided